CLINICAL TRIAL: NCT04936347
Title: A Randomized Controlled Study of Bipolar Electric Cutting and Scissors Under Hysteroscopy in the Treatment of the Intrauterine Adhesion
Brief Title: Hysteroscopic "Hot Knife" and "Cold Knife" in the Treatment of the Intrauterine Adhesion
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Fu Xing Hospital, Capital Medical University (Other)
Responsible Party: Principal Investigator, Xiaowu Huang, Director of department, Fu Xing Hospital, Capital Medical University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Z191100006619058
Record Dates: First submitted 2021-06-18; First posted 2021-06-23 (Actual); Last update posted 2021-09-21 (Actual); Status verified 2021-06

CONDITIONS: Intrauterine Adhesion
MeSH Terms: conditions — Gynatresia | interventions — Conization

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Cold knife (Experimental): The interference of the experimental group is to perform intrauterine adhesiolysis with scissors
  Interventions: Procedure: cold knife
- Hot knife (Other): The interference of the control group is to perform intrauterine adhesiolysis with bipolar electric needle electrode, part of the scar tissue removed by electronic loop when it is necessary.
  Interventions: Procedure: hot knife

INTERVENTIONS:
Procedure: cold knife — Transcervical resection of adhesions is performed with scissors to restore the shape of uterine cavity, promote the regeneration and repair of endometrium, and ultimately improve the reproductive prognosis of patients.
  Arms: Cold knife
Procedure: hot knife — Transcervical resection of adhesions is performed with bipolar electric cutting to restore the shape of uterine cavity, promote the regeneration and repair of endometrium, and ultimately improve the reproductive prognosis of patients.
  Arms: Hot knife

SUMMARY:
In this prospective, randomized controlled trial，the investigators wish to explore the difference of therapeutic effect and prognosis between "hot knife" and "cold knife" in the treatment of uterine adhesion under hysteroscopy.

DETAILED DESCRIPTION:
1. Study Design：This is a prospective, randomized controlled trial.The investigators use hysteroscopy finding as standard reference.
2. Study population 802 patients diagnosed with intrauterine adhesions（IUA）will be prospectively recruited. Before the surgery all patients will undergo preoperative evaluations, including a detailed history of the menstrual pattern,any previous intrauterine surgery, and reproductive history, as well as trans-vaginal ultrasonography.The severity and extent of intrauterine adhesions will be scored according to the ESGE IUA grades.
3. Randomization:

   Randomization was performed electronically using SPSS statistical software version 26.0 (SPSS, Inc., Chicago, IL,USA) by the investigator.802 recruited patients will be randomized to one of the two treatment groups by computer-generated numbers: the control group("hot knife" group) and the experimental group("cold knife" group).
4. Surgical technique:

   * Hysteroscopic surgery will be performed in a standardized manner.The procedure will be performed under general anesthesia. Ultrasonographic guidance will be routinely used.
   * The interference of "cold knife" group (the experimental group) including 401 IUA patients is to perform intrauterine adhesiolysis with scissors, while the interference of "hot knife" group (the control group) is to perform intrauterine adhesiolysis with bipolar electric needle electrode, part of the scar tissue removed by electronic loop when it is necessary.
   * A Foley-catheter filled with 3.0-5.0 ml normal saline will be inserted into the uterus for 5-7 days after surgery.
5. Postoperative treatments

   * All subjects will be treated with oral antibiotics for 5-7 days.
   * All subjects will be treated with Hormone therapy.
   * A second-look hysteroscopy will be carried out in the early proliferative phase 4 weeks after the surgery and an optional third-look hysteroscopy will be carried out 8 weeks after the surgery.
6. Follow up:

   * Follow-up styles: the doctor's outpatient review, telephone, WeChat and so on.
   * Follow-up time:1 month, 2months, 12 months after the operation.
   * Follow up the results of hysteroscopy and the menstrual improvement and pregnancy outcomes at 12 months after the operation.
7. Consent： All subjects will be given a detailed explanation of the study and sufficient time to consider their participation. A written consent form will be signed by the patient and retained in the records.

ELIGIBILITY:
Inclusion Criteria:

* Indications: fertility desire, periodic pelvic pain;
* Women aged 18-40 years;
* Moderate to severe intrauterine adhesion(ESGE Grade II-IV);
* All enrolled women provided written informed consent and agree to the entire study protocol prior to surgery

Exclusion Criteria:

* Contraindications: such as severe medical diseases, pregnancy status, reproductive tract infection, malignant tumor;
* History of uterine artery embolization;
* Infertility caused by male factors or ovarian dysfunction or premature ovarian failure

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 802 (Estimated)
Dates: Start 2019-08-01 (Actual); Primary Completion 2021-12-31 (Estimated); Study Completion 2022-08-31 (Estimated)

PRIMARY OUTCOMES:
Recurrence rate | 2 months after surgery
  Recurrence rate of intrauterine adhesions

SECONDARY OUTCOMES:
Pregnancy rate | 1 year after the patient desire for pregnancy
  The conception rate
Menstrual improvement rate | 2 months after surgery
  The patients' estrual improvement rate

CONTACTS AND LOCATIONS:
Overall Officials: Tinchiu Li, Study Chair — Fuxing Hospital,Capital Medical University
Locations (1):
- Fu Xing Hospital, Capital Medical University, Beijing, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] AAGL Elevating Gynecologic Surgery. AAGL practice report: practice guidelines on intrauterine adhesions developed in collaboration with the European Society of Gynaecological Endoscopy (ESGE). Gynecol Surg. 2017;14(1):6. doi: 10.1186/s10397-017-1007-3. Epub 2017 May 1. No abstract available. PMID 28603474
- [Background] Guo EJ, Chung JPW, Poon LCY, Li TC. Reproductive outcomes after surgical treatment of asherman syndrome: A systematic review. Best Pract Res Clin Obstet Gynaecol. 2019 Aug;59:98-114. doi: 10.1016/j.bpobgyn.2018.12.009. Epub 2019 Jan 3. PMID 30713131
- [Background] Valle RF, Sciarra JJ. Intrauterine adhesions: hysteroscopic diagnosis, classification, treatment, and reproductive outcome. Am J Obstet Gynecol. 1988 Jun;158(6 Pt 1):1459-70. doi: 10.1016/0002-9378(88)90382-1. PMID 3381869
- [Background] Yu D, Wong YM, Cheong Y, Xia E, Li TC. Asherman syndrome--one century later. Fertil Steril. 2008 Apr;89(4):759-79. doi: 10.1016/j.fertnstert.2008.02.096. PMID 18406834
- [Background] Khan Z, Goldberg JM. Hysteroscopic Management of Asherman's Syndrome. J Minim Invasive Gynecol. 2018 Feb;25(2):218-228. doi: 10.1016/j.jmig.2017.09.020. Epub 2017 Oct 9. PMID 29024798
- [Result] Hooker AB, Lemmers M, Thurkow AL, Heymans MW, Opmeer BC, Brolmann HA, Mol BW, Huirne JA. Systematic review and meta-analysis of intrauterine adhesions after miscarriage: prevalence, risk factors and long-term reproductive outcome. Hum Reprod Update. 2014 Mar-Apr;20(2):262-78. doi: 10.1093/humupd/dmt045. Epub 2013 Sep 29. PMID 24082042